CLINICAL TRIAL: NCT01972217
Title: A Randomised, Double-Blind, Placebo-Controlled, Multicentre Phase II Study to Compare the Efficacy, Safety and Tolerability of Olaparib Versus Placebo When Given in Addition to Abiraterone Treatment in Patients With Metastatic Castrate-Resistant Prostate Cancer Who Have Received Prior Chemotherapy Containing Docetaxel
Brief Title: Ph II Study to Evaluate Olaparib With Abiraterone in Treating Metastatic Castration Resistant Prostate Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D081DC00008; UVA97934 (Other: Quintiles); 2013-003520-37 (EudraCT Number)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Olaparib; castration-resistant, metastatic prostate cancer; Prior Docetaxel Chemotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib; abiraterone; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olaparib (Active Comparator): 200 mg or 300 mg bid
  Interventions: Drug: Olaparib; Drug: Abiraterone; Drug: Prednisone or prednisolone
- Placebo (Placebo Comparator): placebo to match olaparib bid
  Interventions: Drug: Placebo; Drug: Abiraterone; Drug: Prednisone or prednisolone

INTERVENTIONS:
Drug: Olaparib — Olaparib bid
  Other Names: PARP inhibition
  Arms: Olaparib
Drug: Placebo — Placebo bid
  Other Names: Placebo to PARP inhibition
  Arms: Placebo
Drug: Abiraterone — Abiraterone 1000 mg
Drug: Prednisone or prednisolone — Prednisone or prednisolone 5 mg bid will be co-administered with the abiraterone in this study.

SUMMARY:
This is a 2-part study in patients with metastatic CRPC. Part A is an open-label safety run-in study to assess the safety, tolerability and pharmacokinetics (PK) of olaparib when given in addition to abiraterone 1000 mg once daily. Part B is a randomised, double-blind, placebo controlled comparison of the efficacy, safety and tolerability of the dose of olaparib selected from Part A when given in addition to abiraterone, versus placebo given in addition to abiraterone. Abiraterone is indicated in combination with prednisone or prednisolone for the treatment of patients with metastatic CRPC. Prednisone or prednisolone 5 mg twice daily (bid) will be administered with the abiraterone in this study.

DETAILED DESCRIPTION:
This is a 2-part study in patients with metastatic CRPC. Part A is an open-label safety run-in study to assess the safety, tolerability and PK of olaparib when given in addition to abiraterone 1000 mg once daily. Part B is a randomised, double-blind, placebo-controlled comparison of the efficacy, safety and tolerability of the dose of olaparib selected from Part A when given in addition to abiraterone, versus placebo in addition to abiraterone.

Abiraterone is indicated in combination with prednisone or prednisolone for the treatment of patients with metastatic CRPC. Prednisone or prednisolone 5 mg bid will be administered with the abiraterone in this study, but throughout this protocol the treatment will be referred to simply as abiraterone.

For Part A of the study, 15 to 18 evaluable patients (Cohorts 1 and 2) are planned to be enrolled from approximately 4 sites in approximately 1 or 2 countries, and a further 12 patients may be recruited into a 3rd cohort if necessary.

For Part B of the study, approximately 140 patients who have received prior chemotherapy containing docetaxel will be randomised from approximately 40 sites in North America and Europe. Patients who have been dosed in Part A of the study may not participate in Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study specific procedures.
2. Male aged 18 years and older.
3. Histologically or cytologically proven diagnosis of prostate cancer.
4. Candidate for abiraterone therapy with documented evidence of metastatic castration-resistant prostate cancer. Metastatic status is defined as at least one documented metastatic lesion on either bone scan or CT/MRI scan. Castration resistant prostate cancer is defined as rising PSA or other signs of disease progression despite treatment with androgen deprivation therapy and the presence of a castrate level of testosterone (≤50 ng/dL).
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2 with no deterioration over the previous 2 weeks.
6. Patients must have a life expectancy ≥12 weeks.
7. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations, and completing PRO instruments.
8. Patients must be on a stable concomitant medication regimen, defined as no changes in medication or in dose within 2 weeks prior to start of olaparib dosing, except for bisphosphonates, denosumab and corticosteroids, which should be stable for at least 4 weeks prior to start of olaparib dosing.
9. For the randomised phase only, patients must have received chemotherapy in the form of docetaxel treatment for metastatic castration-resistant prostate cancer. Note: patients who discontinued docetaxel for toxicity reasons and without completing the full course will still be eligible to enter this study provided they received at least 2 cycles of chemotherapy.

Provide informed consent for the pharmacogenetic sampling and analyses.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff, its agents and/or staff at the study site).
2. Previous treatment in the present study.
3. Treatment with any of the following:

   * Previous exposure to any 2nd generation anti-hormonal including abiraterone and enzalutamide
   * More than 2 prior courses of chemotherapy for metastatic prostate cancer
   * Previous use of immunotherapy or radium-223 for the treatment of metastatic prostate cancer
   * Any investigational agents or study drugs from a previous clinical study within 30 days of the first dose of study treatment;
   * Any previous exposure to a CYP17 (17α-hydroxylase/C17,20-lyase) inhibitor;
   * Substrates of CYP2D6 with a narrow therapeutic index (eg, thioridazine);
   * Potent inhibitors or inducers of CYP3A4 within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort).
   * Any previous treatment with a PARP inhibitor, including olaparib.
4. With the exception of alopecia or toxicities related to the use of gonadotropinreleasing hormone agonists, any unresolved toxicities from prior therapy greater than CTCAE Grade 2 at the time of starting study treatment.
5. Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
6. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
7. Any of the following cardiac criteria:

   * Mean resting QTc >470 msec obtained from 3 ECGs
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval.
8. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years.
9. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count (ANC) <1.5 x 109/L
   * Platelet count <100 x 109/L
   * Haemoglobin (Hb) <100 g/L
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN) if no demonstrable liver metastases or >5 x ULN in the presence of liver metastases
   * Total bilirubin >1.5 x ULN if no liver metastases or >3 x ULN in the presence of liver metastases (except in the case of Gilbert's disease)
   * Creatinine >1.5 x ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 x ULN
   * If bone metastases are present and liver function is otherwise considered adequate by the Investigator then elevated alkaline phosphatase (ALP) will not exclude the patient.
10. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of olaparib or abiraterone.
11. History of hypersensitivity to active or inactive excipients of olaparib or abiraterone or drugs with a similar chemical structure or class to olaparib or abiraterone.
12. Patients with myelodysplastic syndrome/acute myeloid leukaemia.
13. Current disease or condition known to interfere with absorption, distribution, metabolism, or excretion of drugs, at the Investigator's discretion.
14. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
15. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

    Exclusion from the genetic research may be for any of the exclusion criteria specified in the main study or any of the following:
16. Previous allogeneic bone marrow transplant.
17. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the pharmacogenetic sample collection.

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (2):
  - Research Site, San Diego, California
  - Research Site, Lake Success, New York
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Liège
  - Research Site, Wilrijk
- Canada (3):
  - Research Site, London, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Czechia (2):
  - Research Site, Brno
  - Research Site, Liberec
- France (3):
  - Research Site, Angers
  - Research Site, Dijon
  - Research Site, Lyon
- Italy (5):
  - Research Site, Lecce
  - Research Site, Mirano
  - Research Site, Napoli
  - Research Site, Parma
  - Research Site, Pisa
- Netherlands (3):
  - Research Site, Arnhem
  - Research Site, Maastricht
  - Research Site, Nijmegen
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Warsaw
- Russia (3):
  - Research Site, Ivanovo
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Spain (7):
  - Research Site, Badalona
  - Research Site, Córdoba
  - Research Site, Girona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Palma de Mallorca
  - Research Site, Valencia
- United Kingdom (6):
  - Research Site, Cardiff
  - Research Site, Exeter
  - Research Site, Manchester
  - Research Site, Plymouth
  - Research Site, Torquay
  - Research Site, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Clarke N, Wiechno P, Alekseev B, Sala N, Jones R, Kocak I, Chiuri VE, Jassem J, Flechon A, Redfern C, Goessl C, Burgents J, Kozarski R, Hodgson D, Learoyd M, Saad F. Olaparib combined with abiraterone in patients with metastatic castration-resistant prostate cancer: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2018 Jul;19(7):975-986. doi: 10.1016/S1470-2045(18)30365-6. Epub 2018 Jun 4. PMID 29880291
- [Derived] Saad F, Thiery-Vuillemin A, Wiechno P, Alekseev B, Sala N, Jones R, Kocak I, Chiuri VE, Jassem J, Flechon A, Redfern C, Kang J, Burgents J, Gresty C, Degboe A, Clarke NW. Patient-reported outcomes with olaparib plus abiraterone versus placebo plus abiraterone for metastatic castration-resistant prostate cancer: a randomised, double-blind, phase 2 trial. Lancet Oncol. 2022 Oct;23(10):1297-1307. doi: 10.1016/S1470-2045(22)00498-3. Epub 2022 Sep 2. PMID 36063830
- See also: Redacted SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1885&filename=d081dc00008-statistical-analysis-plan-ed-2_Redacted.pdf
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081DC00008&attachmentIdentifier=554eda74-645d-4f7f-afad-0732eb970b3f&fileName=d081dc00008-study-synopsis_(002)_Redacted_27Sep2023.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this 2-part study, patients with metastatic castrate-resistant prostate cancer (mCRPC) were recruited at 41 sites in Europe, Russia and North America. Part A had 2 cohorts for olaparib dose selection when given with approved treatment abiraterone. Part B compared olaparib versus placebo both with abiraterone in post-chemotherapy mCRPC patients.
Pre-assignment Details: Patients dosed in open-label Part A could not participate in Part B which was a randomised, double-blind, placebo-controlled comparison of olaparib + abiraterone versus placebo + abiraterone in patients who had received prior chemotherapy containing docetaxel.
Groups:
- Part A Cohort 1: Olaparib 200 mg + Abiraterone: Patients received olaparib 200 milligrams (mg) twice daily (bid) and abiraterone 1000 mg once daily. Patients were assessed at Weeks 1, 2 and 4, then every 4 weeks up to Week 52, and every 12 weeks thereafter.
  Patients also received prednisone or prednisolone 5 mg bid in combination with the abiraterone treatment.
- Part A Cohort 2: Olaparib 300 mg + Abiraterone: If the combination of olaparib 200 mg + abiraterone 1000 mg was well tolerated (determined after a minimum of 14 days treatment in Cohort 1), patients were recruited into Cohort 2.
  Cohort 2 Group 1: patients received olaparib 300 mg bid alone for 3 to 7 days. Patients then received olaparib 300 mg bid and abiraterone 1000 mg once daily for at least 5 days.
  Cohort 2 Group 2: patients received abiraterone 1000 mg once daily alone for 5 to 7 days. Patients then received olaparib 300 mg bid and abiraterone 1000 mg once daily for at least 3 days.
  Patients also received prednisone or prednisolone 5 mg bid in combination with the abiraterone treatment.
- Part B: Olaparib + Abiraterone: Patients received the selected dose of olaparib 300 mg bid + abiraterone 1000 mg once daily. Patients were assessed every 4 weeks up to Week 52, and every 12 weeks thereafter.
  Patients also received prednisone or prednisolone 5 mg bid in combination with the abiraterone treatment.
- Part B: Placebo + Abiraterone: Patients received placebo bid + abiraterone 1000 mg once daily. Patients were assessed every 4 weeks up to Week 52, and every 12 weeks thereafter.
  Patients also received prednisone or prednisolone 5 mg bid in combination with the abiraterone treatment.
Period: Part A: Open-label Safety Run-in Period
Arm/Group | Part A Cohort 1: Olaparib 200 mg + Abiraterone | Part A Cohort 2: Olaparib 300 mg + Abiraterone | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Started | 3 | 13 | 0 | 0
Completed | 2 | 1 | 0 | 0
Not Completed | 1 | 12 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Condition under investigation worsened | 1 | 9 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Period: Part B Double-blind, Randomised Period
Arm/Group | Part A Cohort 1: Olaparib 200 mg + Abiraterone | Part A Cohort 2: Olaparib 300 mg + Abiraterone | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Started | 0 (Patients recruited to Part A did not participate in Part B.) | 0 (Patients recruited to Part A did not participate in Part B.) | 71 (Patients recruited to Part B did not participate in Part A.) | 71 (Patients recruited to Part B did not participate in Part A.)
Received Olaparib/Placebo | 0 | 0 | 71 | 71
Received Abiraterone | 0 | 0 | 71 | 71
Completed | 0 | 0 | 25 | 24
Not Completed | 0 | 0 | 46 | 47
Not completed — Death | 0 | 0 | 43 | 44
Not completed — Reason not recorded | 0 | 0 | 1 | 0
Not completed — Screen failure | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety analysis set consisted of all patients who received at least 1 dose of study treatment in Part A and all patients randomised into Part B of the study who received at least 1 dose of study treatment.
Groups:
- Part A Cohort 1: Olaparib 200 mg + Abiraterone: Patients received olaparib 200 mg bid and abiraterone 1000 mg once daily. Patients were assessed at Weeks 1, 2 and 4, then every 4 weeks up to Week 52, and every 12 weeks thereafter.
  Patients also received prednisone or prednisolone 5 mg bid in combination with the abiraterone treatment.
- Total: Total of all reporting groups
Arm/Group | Part A Cohort 1: Olaparib 200 mg + Abiraterone | Part A Cohort 2: Olaparib 300 mg + Abiraterone | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone | Total
Number analyzed (Participants) | 3 | 13 | 71 | 71 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 17 | 22 | 42
  >=65 years | 3 | 10 | 54 | 49 | 116
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3 | 13 | 71 | 71 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 11 | 5 | 17
  Not Hispanic or Latino | 2 | 13 | 58 | 63 | 136
  Unknown or Not Reported | 0 | 0 | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 2
  White | 3 | 13 | 67 | 67 | 150
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Patients Experiencing Adverse Events (AEs)
Description: The safety and tolerability of olaparib in combination with abiraterone was assessed during Part A of the study. The percentage of patients experiencing AEs, including information on seriousness, severity, study treatment relationship and those leading to discontinuation for all doses of olaparib and for abiraterone are presented.
  Severity of AEs was assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse events (CTCAE) v4.0. AEs were assigned to a Grade from 1 through 5 as follows:
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life-threatening requiring hospitalisation; Grade 4: Life-threatening consequences; Grade 5: Death related to AE.
  'c-r' = causally related 'discont' = discontinuation.
Time Frame: Cohort 1 and 2: From baseline in Part A (Day 1 for each cohort) up to 30 days following last dose of study treatment.
Population: The Part A Safety analysis set consisted of all patients who received at least 1 dose of study treatment in Part A. Treatment group comparisons were based on the initial dose of olaparib actually received.
Measure: Number; unit: Percentage of patients
Arm/Group | Part A Cohort 1: Olaparib 200 mg + Abiraterone | Part A Cohort 2: Olaparib 300 mg + Abiraterone
Number analyzed (Participants) | 3 | 13
Percentage of patients
  Any AE c-r to olaparib + abiraterone | 66.7 | 46.2
  Any AE c-r to olaparib only | 33.3 | 7.7
  Any AE c-r to abiraterone only | 0 | 15.4
  Any AE CTCAE Grade 3 or higher | 66.7 | 23.1
  Any AE CTCAE Grade 3 or higher c-r to olaparib | 0 | 7.7
  Any AE CTCAE Grade 3 or higher c-r to abiraterone | 0 | 7.7
  Any AE with outcome = death | 0 | 0
  Any serious AE (SAE) | 66.7 | 23.1
  Any SAE c-r to olaparib | 0 | 0
  Any SAE c-r to abiraterone | 0 | 0
  Any AE causing discont of olaparib | 0 | 7.7
  Any AE causing discont of olaparib c-r to olaparib | 0 | 0
  Any AE causing discont olaparib c-r to abiraterone | 0 | 0

2. Primary Outcome: Part A: Number of Patients With Dose Limiting Toxicities (DLTs)
Description: DLTs were assessed by a Safety Review Committee (SRC) after a minimum of 3 patients had received at least 14 days of treatment in Part A.
  A DLT was defined as any toxicity which was not a recognised AE of abiraterone or prednisolone, and was not attributable to the disease or disease-related processes under investigation, which occurred during a minimum period of 14 days treatment and which included: 1. haematological toxicity CTCAE v4.0 Grade 4 or higher present for more than 4 days (except anaemia); 2. non-haematological toxicity CTCAE v4.0 Grade 3 or higher including infection, corrected QT interval prolongation; 3. any other toxicity that was greater than that at baseline, was clinically significant and/or unacceptable, did not respond to supportive care, resulted in a disruption of dosing schedule of 7 days or more, or was judged to be a DLT by the SRC.
  A DLT excluded alopecia and isolated laboratory changes of any grade without clinical sequelae or clinical significance.
Time Frame: From Day 1 for Cohort 1 and from Day 4 for Cohort 2 up to 14 days treatment with olaparib + abiraterone for 3 patients.
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Part A Cohort 1: Olaparib 200 mg + Abiraterone | Part A Cohort 2: Olaparib 300 mg + Abiraterone
Number analyzed (Participants) | 3 | 13
Patients | 2 | 4

3. Primary Outcome: Part B: Median Radiological Progression-Free Survival (rPFS) Time
Description: The efficacy of olaparib when given in combination with abiraterone was assessed by rPFS, defined as the time from randomisation to disease progression using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 (for soft tissue disease) and Prostate Cancer Working Group 2 (PCWG-2) (for bone disease) criteria, or death.
  Progression using RECIST 1.1 criteria was defined as at least 20% increase from baseline in the sum of diameters of target lesions, progression of existing non-target lesions, or the appearance of at least 1 new lesion.
  Progression using PCWG-2 criteria was determined if 2 or more new metastatic bone lesions were observed (with a total of at least 4 new lesions since baseline assessment if observed at the 12 week scan, or persistence of or increase in number of lesions if observed after the 12 week scan as determined by a confirmatory scan at least 6 weeks later or at next scheduled visit).
Time Frame: From baseline, every 12 weeks up to Week 72, then every 24 weeks up to 24 months.
Population: The Full analysis set consisted of all randomised patients in Part B, regardless of treatment actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Months | 13.8 [10.8 to 20.4] | 8.2 [5.5 to 9.7]

4. Primary Outcome: Part B: Percentage of Patients With Progression Events or Death (rPFS)
Description: The efficacy of olaparib when given in combination with abiraterone was assessed by rPFS, defined as the time from randomisation to disease progression using RECIST version 1.1 (for soft tissue disease) and PCWG-2 (for bone disease) criteria, or death.
  Progression using RECIST 1.1 criteria was defined as at least 20% increase from baseline in the sum of diameters of target lesions, progression of existing non-target lesions, or the appearance of at least 1 new lesion.
  Progression using PCWG-2 criteria was determined if 2 or more new metastatic bone lesions were observed (with a total of at least 4 new lesions since baseline assessment if observed at the 12 week scan, or persistence of or increase in number of lesions if observed after the 12 week scan as determined by a confirmatory scan at least 6 weeks later or at next scheduled visit).
  The percentage of patients with progression events is presented overall and according to RECIST 1.1 and/or PCWG-2 criteria, or death.
Time Frame: From baseline, every 12 weeks up to Week 72, then every 24 weeks up to 24 months.
Population: The Full analysis set consisted of all randomised patients in Part B, regardless of treatment actually received.
Measure: Number; unit: Percentage of patients
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Percentage of patients | 64.8 | 76.1
Statistical Analysis 1: Comparison: Part B: Olaparib + Abiraterone vs Part B: Placebo + Abiraterone; The 1-sided p-value provides a test for rejecting the null hypothesis of no treatment effect versus the superiority alternative that patients on olaparib have a lower risk of progression compared with placebo; Test type: Superiority; p = 0.017, Log Rank; Hazard Ratio (HR) = 0.651, 95% CI 2-sided [0.438 to 0.969]

5. Secondary Outcome: Part A Pharmacokinetics (PK): Olaparib Maximum Plasma Concentration at Steady State (Cmax,ss)
Description: Following multiple dosing to steady state of olaparib 300 mg bid, the Cohort 2 olaparib Cmax,ss is presented for olaparib monotherapy and for olaparib given in combination with abiraterone.
  Only patients with data available for analysis at each time point are presented.
Time Frame: PK sampling for Cohort 2 Group 1 was between Days 3 and 7 for olaparib, and Days 4 and 8 for olaparib and abiraterone. PK sampling for Cohort 2 Group 2 was between Days 5 and 7 for abiraterone, and Days 6 and 8 for olaparib and abiraterone.
Population: The PK analysis set consisted of all patients who received at least 1 dose of olaparib per the protocol, for whom there was at least 1 reportable PK concentration and who had no important protocol deviations or AEs that impacted on PK on all PK sampling days. Only patients with data available for analysis at each time point are presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per millilitre (mcg/mL)
Groups:
- Part A Cohort 2 Group 1: Olaparib, Olaparib + Abiraterone: Patients received olaparib 300 mg bid alone for 3 to 7 days to determine the steady state PK profile for olaparib. Patients then received olaparib 300 mg bid and abiraterone 1000 mg once daily for at least 5 days to determine the PK profiles of both olaparib and abiraterone.
  Patients also received prednisone or prednisolone 5 mg bid in combination with the abiraterone treatment.
- Part A Cohort 2 Group 2: Abiraterone, Olaparib + Abiraterone: Patients received abiraterone 1000 mg once daily alone for 5 to 7 days to determine the steady state PK profile for abiraterone. Patients then received olaparib 300 mg bid and abiraterone 1000 mg once daily for at least 3 days to determine the PK profiles of both olaparib and abiraterone.
  Patients also received prednisone or prednisolone 5 mg bid in combination with the abiraterone treatment.
Arm/Group | Part A Cohort 2 Group 1: Olaparib, Olaparib + Abiraterone | Part A Cohort 2 Group 2: Abiraterone, Olaparib + Abiraterone
Number analyzed (Participants) | 7 | 6
micrograms per millilitre (mcg/mL)
  Olaparib alone: number analyzed (Participants) | 6 | 0
  Olaparib alone | 7.781 (25.06) |
  Olaparib + abiraterone: number analyzed (Participants) | 5 | 6
  Olaparib + abiraterone | 6.504 (20.90) | 7.724 (28.05)

6. Secondary Outcome: Part A PK: Abiraterone Cmax,ss
Description: Following multiple dosing to steady state of abiraterone 1000 mg once daily, the Cohort 2 abiraterone Cmax,ss is presented for abiraterone monotherapy and for olaparib given in combination with abiraterone.
  Only patients with data available for analysis at each time point are presented.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Part A Cohort 2 Group 1: Olaparib, Olaparib + Abiraterone | Part A Cohort 2 Group 2: Abiraterone, Olaparib + Abiraterone
Number analyzed (Participants) | 7 | 6
nanograms per millilitre (ng/mL)
  Abiraterone alone: number analyzed (Participants) | 0 | 6
  Abiraterone alone |  | 145.8 (135.5)
  Olaparib + abiraterone: number analyzed (Participants) | 6 | 4
  Olaparib + abiraterone | 130.7 (68.87) | 86.12 (48.88)

7. Secondary Outcome: Part A PK Analysis: Olaparib Time to Reach Maximum Plasma Concentration at Steady State (Tmax,ss)
Description: Following multiple dosing to steady state of olaparib 300 mg bid, the Cohort 2 olaparib tmax,ss is presented for olaparib monotherapy and for olaparib given in combination with abiraterone.
  Only patients with data available for analysis at each time point are presented.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Part A Cohort 2 Group 1: Olaparib, Olaparib + Abiraterone | Part A Cohort 2 Group 2: Abiraterone, Olaparib + Abiraterone
Number analyzed (Participants) | 7 | 6
Hours (h)
  Olaparib alone: number analyzed (Participants) | 6 | 0
  Olaparib alone | 2.000 [1.00 to 2.17] |
  Olaparib + abiraterone: number analyzed (Participants) | 5 | 6
  Olaparib + abiraterone | 2.080 [2.00 to 4.00] | 2.000 [0.500 to 3.02]

8. Secondary Outcome: Part A PK: Abiraterone Tmax,ss
Description: Following multiple dosing to steady state of abiraterone 1000 mg once daily, the Cohort 2 abiraterone tmax,ss is presented for abiraterone monotherapy and for olaparib given in combination with abiraterone.
  Only patients with data available for analysis at each time point are presented.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A Cohort 2 Group 1: Olaparib, Olaparib + Abiraterone | Part A Cohort 2 Group 2: Abiraterone, Olaparib + Abiraterone
Number analyzed (Participants) | 7 | 6
Hours
  Abiraterone alone: number analyzed (Participants) | 0 | 6
  Abiraterone alone |  | 2.525 [1.00 to 3.00]
  Olaparib + abiraterone: number analyzed (Participants) | 6 | 4
  Olaparib + abiraterone | 3.000 [1.08 to 3.00] | 2.500 [2.00 to 3.02]

9. Secondary Outcome: Part A PK Analysis: Olaparib Minimum Plasma Concentration at Steady State (Cmin,ss)
Description: Following multiple dosing to steady state of olaparib 300 mg bid, the Cohort 2 olaparib Cmin,ss is presented for olaparib monotherapy and for olaparib given in combination with abiraterone.
  Only patients with data available for analysis at each time point are presented.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Part A Cohort 2 Group 1: Olaparib, Olaparib + Abiraterone | Part A Cohort 2 Group 2: Abiraterone, Olaparib + Abiraterone
Number analyzed (Participants) | 7 | 6
mcg/mL
  Olaparib alone: number analyzed (Participants) | 6 | 0
  Olaparib alone | 1.264 (46.58) |
  Olaparib + abiraterone: number analyzed (Participants) | 5 | 6
  Olaparib + abiraterone | 0.9170 (31.56) | 1.279 (65.36)

10. Secondary Outcome: Part A PK: Abiraterone Cmin,ss
Description: Following multiple dosing to steady state of abiraterone 1000 mg once daily, the Cohort 2 abiraterone Cmin,ss is presented for abiraterone monotherapy and for olaparib given in combination with abiraterone.
  Only patients with data available for analysis at each time point are presented.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A Cohort 2 Group 1: Olaparib, Olaparib + Abiraterone | Part A Cohort 2 Group 2: Abiraterone, Olaparib + Abiraterone
Number analyzed (Participants) | 7 | 6
ng/mL
  Abiraterone alone: number analyzed (Participants) | 0 | 6
  Abiraterone alone |  | 8.376 (96.52)
  Olaparib + abiraterone: number analyzed (Participants) | 6 | 4
  Olaparib + abiraterone | 7.983 (163.3) | 6.358 (50.96)

11. Secondary Outcome: Part A PK Analysis: Olaparib Area Under the Plasma Concentration-Time Curve at Steady State (AUCss)
Description: Following multiple dosing to steady state of olaparib 300 mg bid, the Cohort 2 olaparib AUCss is presented for olaparib monotherapy and for olaparib given in combination with abiraterone.
  Only patients with data available for analysis at each time point are presented.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*h/mL
Arm/Group | Part A Cohort 2 Group 1: Olaparib, Olaparib + Abiraterone | Part A Cohort 2 Group 2: Abiraterone, Olaparib + Abiraterone
Number analyzed (Participants) | 7 | 6
mcg*h/mL
  Olaparib alone: number analyzed (Participants) | 6 | 0
  Olaparib alone | 45.27 (31.89) |
  Olaparib + abiraterone: number analyzed (Participants) | 5 | 6
  Olaparib + abiraterone | 40.83 (11.47) | 49.51 (37.30)

12. Secondary Outcome: Part A PK: Abiraterone AUCss
Description: Following multiple dosing to steady state of abiraterone 1000 mg once daily, the Cohort 2 abiraterone AUCss is presented for abiraterone monotherapy and for olaparib given in combination with abiraterone.
  Only patients with data available for analysis at each time point are presented.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A Cohort 2 Group 1: Olaparib, Olaparib + Abiraterone | Part A Cohort 2 Group 2: Abiraterone, Olaparib + Abiraterone
Number analyzed (Participants) | 7 | 6
ng*h/mL
  Abiraterone alone: number analyzed (Participants) | 0 | 6
  Abiraterone alone |  | 825.5 (105.5)
  Olaparib + abiraterone: number analyzed (Participants) | 6 | 4
  Olaparib + abiraterone | 718.9 (102.0) | 524.6 (37.65)

13. Secondary Outcome: Part B: Percentage of Patients Experiencing AEs
Description: The safety and tolerability of olaparib when given in combination with abiraterone was assessed during Part B of the study. The percentage of patients experiencing AEs, including information on seriousness, severity, study treatment relationship and those leading to discontinuation for all doses of olaparib and for abiraterone are presented.
  Severity of AEs was assessed using the NCI Common Terminology CTCAE v4.0. AEs were assigned to a Grade from 1 through 5 as follows:
  Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life-threatening requiring hospitalisation; Grade 4: Life-threatening consequences; Grade 5: Death related to AE.
  'c-r' = causally related. 'discont' = discontinuation. 'ola/pla' = olaparib/placebo.
Time Frame: From first dose of study treatment following randomisation in Part B up to 30 days following last dose of study treatment (up to approximately 3 years).
Population: Part B safety analysis set consisted of all patients randomised into Part B of the study who received at least 1 dose of olaparib/placebo.
Measure: Number; unit: Percentage of patients
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Percentage of patients
  Any AE c-r to ola/pla + abiraterone | 45.1 | 12.7
  Any AE c-r to ola/pla only | 18.3 | 9.9
  Any AE c-r to abiraterone only | 1.4 | 7.0
  Any AE CTCAE Grade 3 or higher | 53.5 | 28.2
  Any AE CTCAE Grade 3 or higher c-r to ola/pla | 23.9 | 5.6
  Any AE CTCAE Grade 3 or higher c-r to abiraterone | 16.9 | 1.4
  Any AE with outcome = death | 5.6 | 1.4
  Any AE with outcome = death c-r to ola/pla | 1.4 | 0
  Any AE with outcome = death c-r to abiraterone | 0 | 0
  Any SAE | 35.2 | 19.7
  Any SAE c-r to ola/pla | 9.9 | 1.4
  Any SAE c-r to abiraterone | 5.6 | 0
  Any AE causing discont of ola/pla | 29.6 | 9.9
  Any AE causing discont of treatment c-r to ola/pla | 16.9 | 5.6
  Any AE causing discont treatment c-r abiraterone | 8.5 | 1.4

14. Secondary Outcome: Part B: Median Best Percentage Change From Baseline in Prostate Specific Antigen (PSA) Levels
Description: The best percentage change from baseline in PSA levels was determined to assess the anti-tumour activity of olaparib when given in addition to abiraterone, compared with placebo given in addition to abiraterone.
  The best percentage change was defined as the biggest reduction in PSA level compared with baseline or smallest increase in the absence of a decrease.
Time Frame: From baseline, then every 4 weeks up to Week 52, and then every 12 weeks.
Population: The Full analysis set consisted of all randomised patients in Part B, regardless of treatment actually received. Only patients with data available for analysis are presented.
Measure: Median (Full Range); unit: Percentage change in PSA level
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Percentage change in PSA level | -54.16 [-100.0 to 533.2] | -49.85 [-100.0 to 230.1]

15. Secondary Outcome: Part B: Percentage of Patients With PSA Responses
Description: The percentages of patients with single visit responses and with confirmed responses are presented to assess the anti-tumour activity of olaparib when given in addition to abiraterone, compared with placebo given in addition to abiraterone.
  A single visit response was defined as any post-dose visit PSA level reduced by 50% or more compared with baseline.
  A confirmed response was defined as a reduction in PSA level of 50% or more on 2 consecutive occasions at least 4 weeks apart compared with baseline.
  Patients may have had more than 1 single visit response or confirmed response but were counted once.
Time Frame: From baseline, then every 4 weeks up to Week 24, and then every 12 weeks.
Population: The Full analysis set consisted of all randomised patients in Part B, regardless of treatment actually received.
Measure: Number (80% Confidence Interval); unit: Percentage of patients
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Percentage of patients
  Single visit response | 50.7 [43.10 to 58.31] | 47.9 [40.29 to 55.49]
  Confirmed response | 47.9 [40.29 to 55.49] | 42.3 [34.74 to 49.77]

16. Secondary Outcome: Part B: Median Best Percentage Change From Baseline in Circulating Tumour Cell (CTC) Level
Description: The median best percentage change from baseline in CTC levels was determined to assess the anti-tumour activity of olaparib when given in combination with abiraterone, compared with placebo given in addition to abiraterone.
  The best percentage change was defined as the biggest CTC level reduction compared with baseline or smallest increase in the absence of a decrease.
Time Frame: From baseline, then every 4 weeks up to Week 24, and then every 12 weeks.
Population: as for outcome 14
Measure: Median (Full Range); unit: Percentage change in CTC level
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Percentage change in CTC level | -1.0 [-478 to 613] | -1.0 [-1279 to 414]

17. Secondary Outcome: Part B: Percentage of Patients With at Least One Objective Response (Objective Response Rate [ORR])
Description: The overall radiological ORR was calculated to assess the anti-tumour activity of olaparib in combination with abiraterone, compared with placebo in combination with abiraterone.
  The best overall ORR was defined as the percentage of patients with at least 1 visit response of complete response (CR) or partial response (PR) in soft tissue disease assessed by RECIST 1.1 and also bone scan status of non-progressive disease or non-evaluable for their bone scans assessed by PCWG-2.
  CR: Disappearance of all target lesions. Reduction of pathological lymph nodes to <10 millimetres.
  PR: At least a 30% decrease in the sum of diameters of target lesions from baseline.
  The percentage of patients with a response is presented.
Time Frame: From baseline, then every 4 weeks up to Week 52, and then every 12 weeks.
Population: The Full analysis set consisted of all randomised patients in Part B, regardless of treatment actually received. Only patients with data available for analysis are presented. Only patients with measurable disease at baseline are included.
Measure: Number; unit: Percentage of patients
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Percentage of patients | 27.3 | 31.6
Statistical Analysis 1: Comparison: Part B: Olaparib + Abiraterone vs Part B: Placebo + Abiraterone; Test type: Other; p = 0.309, Regression, Logistic — The p value was calculated with a 1-sided significance level of 2.5%; Odds Ratio (OR) = 0.813, 95% CI 2-sided [0.285 to 2.261]

18. Secondary Outcome: Median Time to First Subsequent Therapy (TFST) and Median Time to Second Subsequent Therapy (TSST)
Description: The TFST and TSST were determined to assess the anti-tumour activity of olaparib when given in combination with abiraterone, compared with placebo given in addition to abiraterone.
  TFST was defined as the time from randomisation to the earlier of first subsequent anti-cancer therapy start date following study treatment discontinuation, or death.
  TSST was defined as the time from randomisation to the earlier of the second subsequent anti-cancer therapy start date following study treatment discontinuation, or death.
Time Frame: From randomisation until analysis cut-off date (up to approximately 3 years).
Population: The Full analysis set consisted of all randomised patients in Part B, regardless of treatment actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Months
  TFST | 13.5 [11.1 to 17.2] | 9.7 [7.3 to 12.9]
  TSST | 19.6 [16.5 to 25.1] | 18.0 [16.9 to 20.6]
Statistical Analysis 1: Comparison: Part B: Olaparib + Abiraterone vs Part B: Placebo + Abiraterone; Olapatib + abiraterone versus placebo + abiraterone: TFST; Test type: Other; p = 0.095, Log Rank — The p value was calculated with a 1-sided significance level of 2.5%; Hazard Ratio (HR) = 0.781, 95% CI 2-sided [0.540 to 1.130]
Statistical Analysis 2: Comparison: Part B: Olaparib + Abiraterone vs Part B: Placebo + Abiraterone; Olaparib + abiraterone versus placebo + abiraterone: TSST; Test type: Other; p = 0.147, Log Rank — The p value was calculated with a 1-sided significance level of 2.5%; Hazard Ratio (HR) = 0.809, 95% CI 2-sided [0.545 to 1.201]

19. Secondary Outcome: Part B: Median Overall Survival (OS)
Description: OS was determined to assess the efficacy of olaparib when given in addition to abiraterone, compared with placebo given in addition to abiraterone.
  OS was performed at the time of the analysis of rPFS, and the median OS, calculated using the Kaplan-Meier technique, is presented.
Time Frame: From baseline, every 12 weeks up to Week 72, then every 24 weeks up to 24 months.
Population: The Full analysis set consisted of all randomised patients in Part B, regardless of treatment actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Months | 22.7 [17.4 to 29.4] | 20.9 [17.6 to 26.3]
Statistical Analysis 1: Comparison: Part B: Olaparib + Abiraterone vs Part B: Placebo + Abiraterone; Test type: Other; p = 0.331, Log Rank — The p value was calculated with a 1-sided significance level of 2.5%; Hazard Ratio (HR) = 0.911, 95% CI 2-sided [0.600 to 1.384]

20. Secondary Outcome: Part B: Median Time to Second Progression or Death (PFS2)
Description: The efficacy of olaparib when given in combination with abiraterone was assessed by PFS2, defined by local standard clinical practice and included objective radiological progression by RECIST 1.1 (soft tissue), symptomatic progression, rise in PSA level or death in the absence of overall progression.
Time Frame: From randomisation until analysis cut-off date (up to approximately 3 years).
Population: The Full analysis set consisted of all randomised patients in Part B, regardless of treatment actually received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
Number analyzed (Participants) | 71 | 71
Months | 23.3 [17.4 to NA] — Insufficient number of patients with events to allow calculation of upper limit for 95% confidence interval. | 18.5 [16.1 to 23.8]
Statistical Analysis 1: Comparison: Part B: Olaparib + Abiraterone vs Part B: Placebo + Abiraterone; Test type: Other; p = 0.140, Log Rank — The p value was calculated with a 1-sided significance level of 2.5%; Hazard Ratio (HR) = 0.788, 95% CI 2-sided [0.511 to 1.215]

ADVERSE EVENTS:
Time Frame: Part A: From baseline (Day 1 for each cohort) up to 30 days following last dose of study treatment. Part B: From first dose of study treatment following randomisation up to 30 days following last dose of study treatment (up to approximately 3 years).
Description: The Part A Safety analysis set consisted of all patients who received at least 1 dose of study treatment in Part A. Part B safety analysis set consisted of all patients randomised into Part B of the study who received at least 1 dose of olaparib/placebo.
Arm/Group | Part A Cohort 1: Olaparib 200 mg + Abiraterone | Part A Cohort 2: Olaparib 300 mg + Abiraterone | Part B: Olaparib + Abiraterone | Part B: Placebo + Abiraterone
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/13 | 43/71 | 45/71
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/13 | 25/71 | 14/71
Other Adverse Events (participants affected / at risk) | 3/3 | 7/13 | 63/71 | 52/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: Olaparib 200 mg + Abiraterone (N=3) | Part A Cohort 2: Olaparib 300 mg + Abiraterone (N=13) | Part B: Olaparib + Abiraterone (N=71) | Part B: Placebo + Abiraterone (N=71)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (7) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Internal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort 1: Olaparib 200 mg + Abiraterone (N=3) | Part A Cohort 2: Olaparib 300 mg + Abiraterone (N=13) | Part B: Olaparib + Abiraterone (N=71) | Part B: Placebo + Abiraterone (N=71)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 18 (23) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 8 (8) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 8 (9) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 17 (19) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 3 (3) | 11 (17) | 8 (11)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (5) | 2 (2) | 27 (42) | 15 (16)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (4) | 2 (3) | 14 (26) | 9 (12)
Asthenia (General disorders) | 0 (0) | 0 (0) | 16 (22) | 10 (11)
Fatigue (General disorders) | 1 (1) | 1 (1) | 15 (16) | 9 (11)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 14 (16) | 8 (8)
Peripheral swelling (General disorders) | 0 (0) | 2 (3) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 10 (11) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 8 (9) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 8 (10) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 5 (5) | 1 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (3) | 1 (1) | 3 (3) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 1 (2) | 2 (3) | 1 (2)
Blood urea increased (Investigations) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine output increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 12 (12) | 5 (5)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (3) | 5 (7) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 8 (8) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 17 (21) | 14 (18)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 11 (12) | 9 (9)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 1 (1) | 5 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (8) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3) | 5 (6) | 4 (4)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 4 (5) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 6 (9) | 5 (7)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Euphoric mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 6 (7) | 2 (2)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 11 (17) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 10 (12) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT01972217/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT01972217/SAP_001.pdf